CLINICAL TRIAL: NCT03681561
Title: Phase I/II Study of Nivolumab in Combination With Ruxolitinib in Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: Nivolumab With Ruxolitinib in Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Veronika Bachanova (Other)
Collaborators: Incyte Corporation (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Veronika Bachanova, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-HEM15-027
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — ruxolitinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I:Ruxolitinib and Nivolumab (Experimental): Participants will receive ruxolitinib at their assigned dose taken orally twice daily on a 28-day cycle combined with nivolumab 480 mg IV administered every 4 weeks (i.e. on Day 1 of a 28-day cycle) until disease progression, unacceptable toxicity, or for a maximum of 2 years.
  Interventions: Drug: Ruxolitinib; Drug: Nivolumab
- Phase II: Ruxolitinib and Nivolumab (Experimental): Participants will receive ruxolitinib at 20mg orally twice daily on a 28-day cycle combined with nivolumab 480 mg IV administered every 4 weeks (i.e. on Day 1 of a 28-day cycle) until disease progression, unacceptable toxicity, or for a maximum of 2 years.
  Interventions: Drug: Ruxolitinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Ruxolitinib — Phase I: Ruxolitinib at assigned dose* twice daily by mouth begin Day 1 and continuing daily until study treatment stop.
  * Dose Levels:
    1. (starting) : 10mg twice daily 2: 15mg twice daily 3: 20mg: twice daily
  Phase II: Ruxolitinib 20mg twice daily by mouth begin Day 1 and continuing daily until study treatment stop.
  Other Names: Jakafi
Drug: Nivolumab — Nivolumab 480 mg IV every 4 weeks (Day 1) Until disease progression, unacceptable toxicity, patient refusal or a maximum of 2 years
  Other Names: Opdivo

SUMMARY:
This is a Phase I/II, multicenter, open-label, dose escalation/dose-expansion study to evaluate the tolerability, safety, and the maximum tolerated dose (MTD) of ruxolitinib when given with fixed dose nivolumab in patients with relapsed or refractory classical Hodgkin lymphoma (cHL).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0, 1 or 2.
* Histologically confirmed diagnosis of classical Hodgkin lymphoma that is relapsed or refractory - historical biopsy at last relapse is acceptable. NOTE: a repeat biopsy is not required for Phase I if the historical biopsy was performed at the most recent relapse, without remission in between. A fresh biopsy is not required for Phase II.
* Presence of radiographically measurable disease (defined as the presence one or more ≥ 1.5 cm lesions, as measured in the longest dimension by PET/CT) within 4 weeks of study registration.
* Prior therapy with check-point inhibitors (nivolumab, pembrolizumab, others) and subsequent progressive disease, stable disease or mixed response
* Failed at least 2 prior therapies including cytotoxic chemotherapy including ABVD or similar, autologous transplantation, brentuximab vedotin, allogenic transplantation without active graft versus host disease Note: Patients who are eligible and willing to undergo autologous transplant should not be enrolled on this trial
* Prior cancer treatment must be completed at least 14 days prior to registration and the patient must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤Grade 1 or baseline. Radiation therapy must be completed at least 7 days prior to registration.
* Absolute Neutrophil Count ≥ 1000/μL
* Platelets ≥ 75,000/μL (or ≥50,000/mm3 if known BM involvement)
* Calculated creatinine clearance ≥ 40 cc/min using the Cockcroft-Gault formula
* Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Males who are sexually active with partners of child-bearing potential must be willing to abstain from heterosexual activity or adhere to contraception from the time of written consent until 7 months after treatment discontinuation.
* Patient must provide voluntary written informed consent prior to the performance of any research related tests or procedures.

Exclusion Criteria:

* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Inability or unwillingness to swallow oral medication or any condition that precludes the administration and/or absorption of oral medications
* A life-threatening illness, medical condition or organ system dysfunction, which in the investigator's opinion, could compromise the patient's safety, interfere with the metabolism of study drugs, or put the study outcomes at undue risk
* Active central nervous system (CNS) involvement by lymphoma
* Uncontrolled cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Concomitant therapy with immunosuppressive agents, including systemic corticosteroids (doses ≤ 10 mg/day prednisone or equivalent are permitted).
* Has a history of autoimmune disease now or in past 3 years such as hepatitis, nephritis, hyperthyroidism, interstitial lung disease or colitis except vitiligo or alopecia, hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
* Active Hepatitis B or C infection (defined as a positive Hepatitis B surface antigen (Ag) or detectable viral load by PCR). NOTES: Hepatitis B and C testing is required. Patients with positive Hepatitis B Ag may enroll if PCR is negative. Suppressive antiviral therapy should be considered for these patients as clinically indicated.
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C
* Currently receiving a strong CYP3A4 Inhibitor (such as but not limited to boceprevir clarithromycin, conivaptan, grapefruit juice, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, voriconazole) or Fluconazole >200 mg/day. Washout period of 1 week is required.
* History of stroke or intracranial hemorrhage within 6 months of study registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 24 months
  To assess the maximum tolerated dose (MTD) of ruxolitinib in combination with nivolumab in patients with relapsed/refractory Hodgkin lymphoma. (Phase I Only)
Overall Disease Control | 24 months
  To evaluate the best Overall Disease Control (CR+PR+SD) at 3 months of nivolumab in combination with ruxolitinib at MTD in patients with relapsed/refractory Hodgkin lymphoma using the modified Lugano Classification "lymphoma response criteria to immunomodulatory therapy criteria" (LYRIC)1 (Phase II Only)

SECONDARY OUTCOMES:
Overall Response Rate | 24 months
  To characterize the Best Overall Response Rate (CR+PR) at 6 months of nivolumab in combination with ruxolitinib in patients with relapsed/refractory classical Hodgkin lymphoma (cHL).
Progression Free Survival | 24 months
  To evaluate progression free survival (PFS) at 2 years for nivolumab in combination with ruxolitinib in patients with relapsed/refractory Hodgkin lymphoma using the modified Lugano Classification "lymphoma response criteria to immunomodulatory therapy criteria" (LYRIC)
Duration of Response | 24 months
  To evaluate duration of response (DOR) at 2 years for nivolumab in combination with ruxolitinib in patients with relapsed/refractory Hodgkin lymphoma using the modified Lugano Classification "lymphoma response criteria to immunomodulatory therapy criteria" (LYRIC)
Overall Survival | 24 months
  To evaluate overall survival (OS) at 2 years for nivolumab in combination with ruxolitinib in patients with relapsed/refractory Hodgkin lymphoma using the modified Lugano Classification "lymphoma response criteria to immunomodulatory therapy criteria" (LYRIC)
Frequency and Severity of Adverse Events as assessed by CTCAE v4.0 | 24 months
  To characterize he safety and tolerability of nivolumab in combination with ruxolitinib as determined by the frequency and severity of adverse events (AEs) as defined by the NCI's Common Terminology Criteria for Adverse Events version 4 (CTCAE v4)

CONTACTS AND LOCATIONS:
Overall Officials: Veronkia Bachanova, Principal Investigator — University of Minnesota
Locations (6):
- United States (6):
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No